CLINICAL TRIAL: NCT04940169
Title: Prospective Comparison Of Arthroscopic Anterior Cruciate Ligament Reconstrictions Made With Hamstring Tendon And Quadriceps Tendon Autografts
Brief Title: Anterior Cruciate Ligament Reconstruction Made With Hamstring Tendon And Quadriceps Tendon Autografts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SB Istanbul Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Neset Tang, attendant, SB Istanbul Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IER Hospital
Record Dates: First submitted 2021-06-11; First posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- quadriceps tendon autograft (Experimental): Ramdomized half of the patient underwent quadriceps graft harvesting. Arthroscopic technique fixation methods rehabilitation style follow periods kept same as hamstring group except graft type.
  Interventions: Procedure: anterior cruciate ligament recontruction
- hamstring tendon autograft (Experimental): Ramdomized half of the patient underwent hamstring graft harvesting. Arthroscopic technique fixation methods rehabilitation style follow periods kept same as hamstring group except graft type.
  Interventions: Procedure: anterior cruciate ligament recontruction

INTERVENTIONS:
Procedure: anterior cruciate ligament recontruction — Firstly graft is harvested with help of arthroscopy femoral and tibial tunnels created then graft placed into tunnels

SUMMARY:
Anterior cruciate ligament reconstruction (ACLR) is one of the most common procedure all around the world, however optimal graft source for ACLR still remains controversial. Although Quadriceps tendon (QT) is the least used and least studied autograft, it could be an appropriate and good alternative for ACLR. If investigaters use the same surgical technique, and exert the same rehabilitation methods they may have better results than hamstring tendon (HT) autografts.

DETAILED DESCRIPTION:
Investigators enrolled 36 patient and randomized them to different group (HT, QT). at the first evaluation examination findings noted, PROMs (patient reported outcome measurements) questioned, thigh circumference measured, flexor and extensor thigh muscle strength recorded with help of Humac CYBEX Norm (CSMI, 2004) device. After these examinations and preparations all patients operated by the same surgeon who is familiar with both technique. The same surgical technique and fixation method used for both groups. At 1st year follow-up all evaluations PROMs (İKDC,lysholm,VAS) and measurements repeated. Back to the sports rates and postoperative complications compared between HT-QT.

ELIGIBILITY:
Inclusion Criteria:

diagnosed primary ACL rupture willing to involve study

* lesser than Outerbridge 2 cartilage lesions, non-buckethandle meniscus injuries

Exclusion Criteria:

more than one ligament injury greater than outerbridge 3 cartilage injury buckethandle meniscus injuries re-ruptures bilateral injuries previous knee surgery any disease affecting muscle strength

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2018-07-06 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
KOOS | Change from Baseline score at one year.
  Simple patient reported questionnaire
lysholm | Change from Baseline score at one year.
  Simple patient reported questionnaire
VAS | Change from baseline score at one year.
  Simple patient reported questionnaire
IKDC | Change from baseline score at one year.
  Simple patient reported questionnaire
STRENGTH TEST | Change from baseline score at one year.
  Simple patient reported questionnaire
subjective instability test | Change from baseline score at one year.
  instability measure with help of examinations
thigh circumference | Change from baseline score at one year.
  circumference measure
one leg hop test | Change from baseline score at one year.
  ask to participant hop on operated leg

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul education and research hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No